CLINICAL TRIAL: NCT03030937
Title: A Randomized, Parallel Control, Exploratory Trial to Compare Apatinib Plus Irinotecan Versus Single Irinotecan as Second-line Treatment in Subjects With Advanced Gastric Cancer or Adenocarcinoma of Esophagogastric Junction
Brief Title: Clinical Trial to Compare Apatinib Plus Irinotecan Versus Single Irinotecan as Second-line Treatment in AGC or EGJA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-G201
Record Dates: First submitted 2017-01-15; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Gastric Cancer Adenocarcinoma of Esophagogastric Junction
MeSH Terms: interventions — apatinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan plus apatinib (Experimental): Irinotecan:160mg/m2, ivgtt,given on the eighth day; Apatinib:initial dose:250mg,oral,once a day, after meal ( try to take the medicine at the same time of the dauntoy ).
  Repeat the therapeutic schedule every 2 weeks till progressive disease or intolerable toxicities.
  Interventions: Drug: Apatinib; Drug: Irinotecan
- Irinotecan (Active Comparator): Irinotecan:180mg/m2, ivgtt,given on the eighth day. Repeat the therapeutic schedule every 2 weeks till progressive disease or intolerable toxicities.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Apatinib — Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2).
  Arms: Irinotecan plus apatinib
Drug: Irinotecan — Irinotecan was used as second line treatment with AGC.

SUMMARY:
The purpose of this study is to determine whether apatinib plus irinotecan can improve progression free survival compared with single irinotecan in patients with advanced gastric cancer or adenocarcinoma of esophagogastric junction who failed one lines of chemotherapy.

DETAILED DESCRIPTION:
Gastric cancer is the leading cause of cancer death in China. Most patients are unresectable or metastatic disease at the time of diagnosis,so the prognosis is poor.Systemic therapy was required for the patients with advanced stage. Platinum combined with fluoropyrimidines always were considered as first line treatment. After failure of initial therapy, single agent of irinotecan was used as second line treatment,but limited survival benefit.Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2).The purpose of this study is to determine whether apatinib plus irinotecan can improve progression free survival compared with single irinotecan in patients with advanced gastric cancer or adenocarcinoma of esophagogastric junction who failed one lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~70years;
2. Subjects with Histologically or cytologically confirmed advanced gastric cancer or adenocarcinoma of esophagogastric junction ；
3. Subjects must have received no more than one lines treatment before participating,and have received no irinotecan or antiangiogenic（including apatinib）treatment previously; Note：(1) Time of first-line treatment for subjects with advanced tumour must more than 1 cycles;(2) Adjuvant / neoadjuvant therapy was allowed; adjuvant / neoadjuvant therapy will be considered as a first-line treatment if disease recurrence during treatment or after less than 24 weeks.
4. subjects with at least one measurable lesion as defined by RECIST (version 1.1);Lesions previously treated with radiotherapy or locoregional therapy must show radiographic evidence of disease progression to be deemed a target lesion.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
6. Survival expectation≥ 3 months;
7. The interval of subjects had received cytotoxic drugs, radiotherapy or surgery must more than 4 weeks(besides nitroso or mitomycin must more than 6 weeks), and the wound has healed before participating;
8. No serious concomitant diseases(including heart,lung,liver jaundice or gastrointestinal obstruction and so on );
9. Adequate organ functions defined as indicated below： （1）Adequate bone marrow function, defined as: (no blood transfusion within 14 days)

   1. Hemoglobin (Hb)≥80g/L，
   2. White blood count (WBC)≥3.5×109/L
   3. Absolute neutrophil count (ANC)≥1.5×109/L，
   4. Platelet count (PLT)≥75×109/L； （2）Adequate liver function, defined as:

   <!-- -->

   1. Bilirubin ≤1.5×the upper limit of normal (ULN)
   2. Alanine aminotransferase (ALT), or Aspartate aminotransferase (AST) ≤3.0×(ULN), Glutamyl transpeptidase(GGT)≤2.5×(ULN), (When liver metastases, ALT or AST and GPT <5.0×(ULN)).
   3. serum creatinine ≤1.0×（ULN）, or creatinine clearance > 50 mL/min( calculated per the Cockcroft and Gault formula)
10. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative, Females of childbearing potential must agree to use a highly effective method of contraception throughout the entire study period and for 8 weeks after study drug discontinuation. Male subjects must have had a successful vasectomy or they and their female partners must meet the criteria above (i.e.not of childbearing potential or practicing highly effective contraception throughout the study period and for 8 weeks after study drug discontinuation).
11. Subjects provided written informed consent before participating,Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Females are lactating or pregnant at Screening or Baseline
2. Subjects with other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix)
3. Subjects with symptomatic brain metastases；
4. Subjects with uncontrolled blood pressure with medication (140/90 mmHg),
5. Subjects with coronary heart disease (CHD) above grade I, arrhythmia (including Prolongation of QTc interval : Male subjects > 450 ms, Females> 470 ms) or cardiac dysfunction;.
6. Subjects with gastrointestinal bleeding tendency,including the following: current of local active ulcerative lesions with fstool OB (+ +); history of melena or hematemesis within past 2 months ; current of fstool OB (+) with gastric primary tumor without surgical , investigator considerd ulcerative stomach cancer is associated with risks of gastrointestinal bleeding.
7. Subjects with bleeding tendency ，defined as abnormal coagulation (INR>1.5×(ULN),APTT>1.5 ×(ULN));
8. Subjects with previous history of cardiovascular and cerebrovascular diseases ,those receiving thrombolytics or anticoagulants were excluded
9. Subjects with urine protein positive (defined as urine protein detection 2+ or above, or urine protein ≥ 1 g/24 hours );
10. Subjects with a variety of factors that affect oral medications (such as inability to swallow, persistent nausea and vomiting, chronic diarrhea and intestinal obstruction, and so on.);
11. Subject with any other condition that in the opinion of the investigator would preclude his/her participation in a clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 18 months
Adverse Event（AE） | 18 months
  NCI CTC 4.03

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 18 months
Disease Control Rate (DCR) | 18 months
Overall Survival(OS) | 18 months
Quality of Life (QoL) | 18 months
  Use the validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 [EORTC QLQ-C30].

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Yang, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Jianwei Yang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided